CLINICAL TRIAL: NCT03317431
Title: the Mechanism of the Downregulation of Dopamine Receptor in Mechanical Ventilation Induced Lung Injury
Brief Title: the Effect of Dopamine on Mechanical Ventilation Induced Lung Injury
Status: Completed | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-17-011
Record Dates: First submitted 2017-07-17; First posted 2017-10-23 (Actual); Results first posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2017-03

CONDITIONS: Acute Lung Injury
Keywords: dopamine,mechanical ventilation,lung injury
MeSH Terms: conditions — Acute Lung Injury | interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Gather the lung tissues from patients undergo lobectomy with general anesthesia and mechanical ventilation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ventilation: patients undergoing selective operation with general anesthesia(GA) and mechanical ventilation(MV)
  Interventions: Other: mechanical ventilation

INTERVENTIONS:
Other: mechanical ventilation — mechanical ventilation protocol: tidal volume 6-8 ml/kg, positive end-expiratory pressure 5 cmH2O, oxygen concentration 40%; respiratory rate 10-15/min, inspiratory/expiratory ratio 1:1.5.

SUMMARY:
Dopamine(DA) is a common neurotransmitter that has been known to regulate behavior, movement, cardiovascular，endocrine and gastrointestinal functions, but also functions as an important molecule engaging in the immune systems to possess anti-inflammatory effects. However, its role in ventilator-induced lung injury (VILI) is still unclear. Herein, this study aimed to investigate the therapeutic efficacy of dopamine on ventilation-induced lung endothelial barrier dysfunction and explore the possible underlying molecular mechanisms.

DETAILED DESCRIPTION:
Mechanical ventilation is a critical intervention for patients with acute respiratory failure. However, lung overdistension induced by mechanical ventilation at high tidal volumes also causes pulmonary endothelial dysfunction. The injurious effect of mechanical stretch on pulmonary endothelium has been implicated in the development of ventilator-induced lung injury (VILI), which is characterized by pulmonary inflammation and particularly increased vascular permeability. In addition, the investigators and others have previously shown that mechanical stretch increases cultured lung endothelial monolayer permeability in vitro and promotes lung vascular permeability in mice Thus, elucidating the mechanisms underlying the mechanical stretch-induced lung endothelial barrier dysfunction may provide a novel clinical therapeutic target against VILI.

Dopamine is a neurotransmitter, which can also be produced outside the central nervous system. Lung alveolar epithelial cells represent an important source of extraneuronal dopamine, which has a significant role in local organ physiology. Dopamine D1 receptor (DRD1) and D2 receptor (DRD2) are present in lung tissues. Activation of D2DR induces NaKATPase gene expression. Moreover, activation of DRD1 results in the trafficking of NaKATPase to the basolateral membrane of type II alveolar epithelial cells, thus increasing lung liquid clearance during acute lung injury. Although the lung-protective effects of DA and its implication in the pathology of ALI are emerging, the mechanisms are still largely unknown.

In the present study, the investigators will analyze the influence of mechanical ventilation on dopamine receptors in the lung tissue of the participants, and explore whether DA could protect ventilation induced lung injury, which is helpful for prevention and treatment of ventilation induced lung injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients inclusion criteria: undergo elective lobectomy with general anesthesia and mechanical ventilation; classified as physical status I to III according to the American Society of Anesthesiologists Physical Status Classification System; Written informed consent is approved.

Exclusion Criteria:

* Distant metastases: recent anaesthetics or mechanical ventilation treatment；children；women during pregnancy or lactation; being involved in other clinical subjects.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients undergo elective lobectom
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-10-22 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lai Jiang, chief doctor, Study Chair — Xinhua Hospital affiliated to Medicine school,Shanghai Jiaotong University
Locations (1):
- Department of Anesthesia, Shanghai Xinhua hospital, Shanghai, Shanghai Municipality, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ventilation
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ventilation
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 46
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 46
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 46

OUTCOME MEASURES:

1. Primary Outcome: Correlation Coefficient (r) Between Duration of Mechanical Ventilation and DRD1 Expression
Description: ImageJ software were used to get the Integrated Optical Density(IOD) of the chemiluminescent signal from the membranes of dopamine receptor 1(DRD1). The normalization was carried out by DRD1 IOD/total β-actin IOD for sample loading correction. In determination of the expression level of DRD1 in different time points, the investigators had a bulk preparation of normal placental protein which was set as a control. Analyze the correlation between duration of mechanical ventilation and DRD1 expression. If p value is less than 0.05, then its change is statically significant.
Time Frame: 20min-60min
Measure: Number; unit: pearson Correlation Coefficient
Arm/Group | Ventilation
Number analyzed (Participants) | 46
pearson Correlation Coefficient | -0.555
Statistical Analysis 1: Comparison: Ventilation; Analysis the relationship between the duration of mechanical ventilation with DRD1 expression; Test type: Superiority; p < 0.01, Regression, Linear

2. Secondary Outcome: Correlation Coefficient (r) Between Duration of Mechanical Ventilation and DRD2 Expression
Description: ImageJ software were used to get the Integrated Optical Density(IOD) of the chemiluminescent signal from the membranes of dopamine receptor 2(DRD2). The normalization was carried out by DRD2 IOD/total β-actin IOD for sample loading correction. In determination of the expression level of DRD2 in different time points, the investigators had a bulk preparation of normal placental protein which was set as a control. Analyze the correlation between duration of mechanical ventilation and DRD2 expression. If p value is less than 0.05, then its change is statically significant.
Time Frame: 20min-60min
Measure: Number; unit: pearson Correlation coefficient
Arm/Group | Ventilation
Number analyzed (Participants) | 46
pearson Correlation coefficient | 0.094
Statistical Analysis 1: Comparison: Ventilation; Analysis the relationship between the duration of mechanical ventilation with DRD2 expression; Test type: Superiority; p > 0.01, Regression, Linear

3. Secondary Outcome: the Expression of TH in Lung Tissues
Description: ImageJ software were used to get the Integrated Optical Density(IOD) of the chemiluminescent signal from the membranes of Tyrosine hydroxylase(TH). The normalization was carried out by TH IOD/total β-actin IOD for sample loading correction. In determination of the expression level of TH in different time points, the investigators had a bulk preparation of normal placental protein which was set as a control. Analyze the correlation between duration of mechanical ventilation and TH expression. If p value is less than 0.05, then its change is statically significant.
Time Frame: 20min-60min
Measure: Number; unit: pearson correlation coefficient
Arm/Group | Ventilation
Number analyzed (Participants) | 46
pearson correlation coefficient | -0.047
Statistical Analysis 1: Comparison: Ventilation; Analysis the relationship between the duration of mechanical ventilation with TH expression; Test type: Superiority; p > 0.01, Regression, Linear

4. Secondary Outcome: the Expression of DDC in Lung Tissues
Description: ImageJ software were used to get the Integrated Optical Density(IOD) of the chemiluminescent signal from the membranes of Dopa decarboxylase(DDC). The normalization was carried out by DDC IOD/total β-actin IOD for sample loading correction. In determination of the expression level of DDC in different time points, the investigators had a bulk preparation of normal placental protein which was set as a control. Analyze the correlation between duration of mechanical ventilation and DDC expression. If p value is less than 0.05, then its change is statically significant.
Time Frame: 20min-60min
Measure: Number; unit: pearson correlation coefficient
Arm/Group | Ventilation
Number analyzed (Participants) | 46
pearson correlation coefficient | -0.012
Statistical Analysis 1: Comparison: Ventilation; Analysis the relationship between the duration of mechanical ventilation with DDC expression; Test type: Superiority; p > 0.01, Regression, Linear

5. Secondary Outcome: the Expression of Ac-a-tubulin in Lung Tissues
Description: ImageJ software were used to get the Integrated Optical Density(IOD) of the chemiluminescent signal from the membranes of acetylated-a-tubulin(Ac-a-tubulin). The normalization was carried out by Ac-a-tubulin IOD/total β-actin IOD for sample loading correction. In determination of the expression level of Ac-a-tubulin in different time points, the investigators had a bulk preparation of normal placental protein which was set as a control. Analyze the correlation between duration of mechanical ventilation and Ac-a-tubulin expression. If p value is less than 0.05, then its change is statically significant.
Time Frame: 20min-60min
Measure: Number; unit: pearson correlation coefficient
Arm/Group | Ventilation
Number analyzed (Participants) | 46
pearson correlation coefficient | -0.465
Statistical Analysis 1: Comparison: Ventilation; Analysis the relationship between the duration of mechanical ventilation with Ac-a-tubulin expression; Test type: Superiority; p < 0.01, Regression, Linear

ADVERSE EVENTS:
Time Frame: 20-60 min
Description: All-Cause Mortality, Serious, and Other Adverse Events were not monitored/assessed.Because the investigators gain the lung tissue from the pathology department after the surgery.
Arm/Group | Ventilation
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT03317431/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT03317431/Prot_SAP_001.pdf